CLINICAL TRIAL: NCT04642586
Title: Detection of Subclinical Cerebral Suffering Related to Hypertension Using Multimodal MRI (SOUCHY) Brain Changes Due to Hypertension: a Multimodal MRI
Brief Title: Detection of Subclinical Cerebral Suffering Related to Hypertension Using Multimodal MRI
Acronym: SOUCHY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC31/19/0055
Record Dates: First submitted 2020-11-06; First posted 2020-11-24 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
Keywords: MRI, Hypertension
MeSH Terms: conditions — Hypertension | interventions — Hematologic Tests

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertensive participants (Experimental): diagnosed HTA within 5 years, treated or confirmed by Ambulatory Blood Pressure Measure;
  Interventions: Diagnostic Test: multimodal magnetic resonance imaging; Diagnostic Test: blood test; Diagnostic Test: neuropsychological assessment
- Normotensive participants (Experimental): absence of HTA confirmed by Ambulatory Blood Pressure Measure
  Interventions: Diagnostic Test: multimodal magnetic resonance imaging; Diagnostic Test: blood test; Diagnostic Test: neuropsychological assessment

INTERVENTIONS:
Diagnostic Test: multimodal magnetic resonance imaging — Brain MRI exam (without contrast injection)
  Other Names: MRI
Diagnostic Test: blood test — Blood test to evaluate cardiovascular risk factors (cholesterol, triglycerides, LDL and HDL-CT, serum creatinine, fasting glucose, serum potassium), .
Diagnostic Test: neuropsychological assessment — neuropsychological assessment

SUMMARY:
Investigators propose here to study the brain consequences of hypertension in patients without cognitive complaints and neurological signs. The evaluation of brain suffering requires considering various possible brain damage. The team developed a multimodal MRI approach capable of detecting and quantifying numerous indices (e.g. morphometric, microstructural) to evaluate possible brain suffering. This project aims to identify individually signs of cerebral suffering in hypertensive patients compared to a population of normotensive volunteers, using advanced multiparametric MRI methods.

DETAILED DESCRIPTION:
Hypertension is a risk factor for many brain pathologies, such as ischemic and hemorrhagic neurodegenerative diseases or stroke. The literature seems to agree on the relationship between hypertension and brain damage, and on the benefit of the management of hypertension to prevent certain neurological pathologies. However, to our knowledge, no single study has shown signs of subclinical brain damage in patients with hypertension. At present, no brain MRI is recommended in these patients. In the present study, hypertensive and normotensive patients will undergo a neurological exam, a neuropsychological exam, a biological exam and a MRI exam to individually identify signs of cerebral suffering.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 35 to 50 y.o.;for patients: diagnosed HTA within 5 years, treated or confirmed by Ambulatory Blood Pressure Measure;
* For normotensive participants:Absence of HTA confirmed by Ambulatory Blood Pressure Measure

Exclusion Criteria:

* Known neurological history, stroke, symptomatic headache, long-term use of neuroleptic, tricyclic, MAOI, anti-serotonergic antidepressant medications, diabetes mellitus, treated dyslipidemia, body mass index greater than 30 kg / m, participants who smoked or smoked more than 10 packs-year, MRI contraindication ;
* For HTA patients only: Renal artery dysplasia responsible for hypertension, clinical Cushing Syndrome.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2023-12-05 (Estimated); Study Completion 2024-01-05 (Estimated)

PRIMARY OUTCOMES:
Presence of a cerebral zone with a z-score > 1.96 | through study completion, an average of 1 year
  the proportion of hypertensive patients who have at least one sign of cerebral suffering compared to the control group will be determined. For each MRI parameter, after coregistration, z score maps will be calculated for each hypertensive patient (individual vs normotensive group). The notion of cerebral suffering sign will be defined by the presence of a cerebral zone with a z-score greater than 1.96 (corresponding to a threshold of significance p <.05).

SECONDARY OUTCOMES:
White matter hypersignals | through study completion, an average of 1 year
  FAZEKAS score estimating T2 hypersignals of the white matter,
Microbleeds | through study completion, an average of 1 year
  number and location of microbleeds,
Gaps | through study completion, an average of 1 year
  number of gaps

OTHER OUTCOMES:
Correlation between MRI data and clinical scales | through study completion, an average of 1 year
  MRI parameters will be correlated with clinical and neuropsychological using Spearman 'rank correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Darcourt, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No